CLINICAL TRIAL: NCT01609075
Title: Use of Bevacizumab in the Treatment of Metastatic Colorectal Cancer (mCRC) in Italy: an Observational Cohort Study
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Colorectal Cancer in Italy (BEWARE)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML27907
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational, multicenter, retrospective/prospective study will evaluate the use of Avastin (bevacizumab) in clinical practice in patients with metastatic colorectal cancer. Patients having initiated first-line treatment with a fluoropyrimidine-based chemotherapy and Avastin will be followed for up to 15 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Metastatic colorectal cancer
* Having initiated first-line treatment with fluoropyrimidine-based chemotherapy plus Avastin between 1. September 2011 and 29. February 2012
* Availability of test fro K-RAS genotyping

Exclusion Criteria:

* Participation in a clinical trial during treatment with Avastin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic colorectal cancer having initiated first-line treatment with fluoropyrimidine-based chemotherapy and Avastin
Sampling Method: Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Avastin treatment discontinuation due to either disease progression or Avastin-related adverse events | approximately 15 months

SECONDARY OUTCOMES:
Proportion of patients with treatment discontinuation due to other causes | approximately 15 months
Incidence of other causes for treatment discontinuation | approximately 15 months
Second-line treatments initiated | approximately 15 months
Progression-free survival (patients with treatment discontinuation due to disease progression or Avastin-related toxicity as compared to patients with treatment discontinuation due to other causes) | approximately 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (65):
- Italy (65):
  - L’Aquila, Abruzzo
  - Teramo, Abruzzo
  - Brindisi, Apulia
  - Castellana Grotte (BA), Apulia
  - Foggia, Apulia
  - Lecce, Apulia
  - San Giovanni Rotondo, Apulia
  - Rionero in Vulture, Basilicate
  - Cosenza, Calabria
  - Lamezia Terme (CZ), Calabria
  - Reggio Calabria, Calabria
  - Benevento, Campania
  - Napoli, Campania
  - Pagani ( Sa), Campania
  - Imola (BO), Emilia-Romagna
  - Modena, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Pordenone, Friuli Venezia Giulia
  - Albano Laziale, Lazio
  - Rome, Lazio
  - Sora, Lazio
  - Viterbo, Lazio
  - Genoa, Liguria
  - La Spezia, Liguria
  - Savona, Liguria
  - Bergamo, Lombardy
  - Brescia, Lombardy
  - Cremona, Lombardy
  - Lecco, Lombardy
  - Milan, Lombardy
  - Monza, Lombardy
  - Pavia, Lombardy
  - S. Fermo Della Battaglia (CO), Lombardy
  - Saronno, Lombardy
  - Varese, Lombardy
  - Cuneo, Piedmont
  - Novara, Piedmont
  - Orbassano, Piedmont
  - Ponderano (BI), Piedmont
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Sassari, Sardinia
  - Catania, Sicily
  - Cefalù, Sicily
  - Messina, Sicily
  - Palermo, Sicily
  - Taormina, Sicily
  - Vimercate, Sicily
  - Fano, The Marches
  - Fermo, The Marches
  - Macerata, The Marches
  - Grosseto, Tuscany
  - Lido di Camaiore, Tuscany
  - Livorno, Tuscany
  - Pontedera, Tuscany
  - Siena, Tuscany
  - Perugia, Umbria
  - Cona (Ferrara), Veneto
  - Este, Veneto
  - Este (PD), Veneto
  - Mirano, Veneto
  - Montecchio Maggiore, Veneto
  - Padua, Veneto
  - Rovigo, Veneto
  - Treviso, Veneto

REFERENCES:
- [Derived] Lonardi S, Nasti G, Fagnani D, Gemma D, Ciuffreda L, Granetto C, Lucchesi S, Ballestrero A, Biglietto M, Proserpio I, Bergamo F, Proietti E, Tonini G. Discontinuation of first-line bevacizumab in metastatic colorectal cancer: the BEAWARE Italian Observational Study. Tumori. 2019 Jun;105(3):243-252. doi: 10.1177/0300891619834126. Epub 2019 Mar 11. PMID 30857495